CLINICAL TRIAL: NCT06206811
Title: A Four-part, Phase 1, Double-blind Study to Investigate the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) with Single and Multiple Ascending Oral Doses of OD-07656 in Healthy, Adult Male and Female Participants
Brief Title: Phase 1 Study to Investigate OD-07656 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Odyssey Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OD-07656-001
Record Dates: First submitted 2023-12-20; First posted 2024-01-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Bowel Diseases; Blau Syndrome; Crohn Disease; Ulcerative Colitis; Spondyloarthritis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Blau syndrome; Crohn Disease; Colitis, Ulcerative; Spondylarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1 - Single Ascending dose (Experimental): To assess the safety and tolerability of single ascending doses of OD-07656 administered as an oral capsule
  Interventions: Drug: OD-07656
- Part 2 - Multiple Ascending dose (Experimental): To assess the safety and tolerability of multiple ascending doses of OD-07656 administered as an oral capsule
  Interventions: Drug: OD-07656
- Part 3 - Food effect and relative bioavailability between dose forms (Experimental): To assess the safety and tolerability of OD-07656 administered as an oral capsule or tablet
  Interventions: Drug: OD-07656
- Part 4 - Pharmacokinetic drug interaction between midazolam and OD-07656 (Experimental): To assess the safety and tolerability of OD-07656 administered as an oral capsule or tablet following administration of midazolam
  Interventions: Drug: OD-07656

INTERVENTIONS:
Drug: OD-07656 — innate immune modulator

SUMMARY:
First-in-human study to provide an assessment of the safety, tolerability, pharmacokinetics (PK), including food effects and a drug-drug interaction, and pharmacodynamics (PD) of OD-07656 after administration of ascending single and multiple oral doses to healthy male and female participants in view of treating inflammatory bowel disease (IBD) (including Crohn's disease and ulcerative colitis), Blau syndrome, and spondyloarthritis

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
2. Body Mass Index (BMI) within the range 18-32kg/m2 (inclusive)
3. Female participants must be of nonchildbearing potential, defined as either surgically sterile (i.e., hysterectomy, bilateral salpingectomy, tubal ligation, or bilateral oophorectomy), OR be post-menopausal with at least 1 year of amenorrhea. Female participants must use barrier contraception to protect against the transfer of study drug in any body fluids from time of first dose and for at least 7 days after the last dose of study drug.
4. Male participants must agree to use double barrier contraception (i.e. a condom and additional contraception for their female partner) when sexually active with a female partner of child-bearing potential from Screening until at least 90 days after the last dose of study drug (or be surgically sterile [i.e., vasectomy with documentation]); or remain abstinent from heterosexual intercourse [when this is in line with the preferred and usual lifestyle] from the time of admission to the clinical centre up to 90 days post last dose. Male participants should also agree not to donate sperm for the duration of the study and until at least 90 days after the last dose of study drug.
5. Male participants who engage in intercourse with same sex partners are required to use barrier forms of contraception to protect against the transfer of study drug in any body fluids from time of first dose and for at least 7 days after the last dose of study drug.
6. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

1. Females with child-bearing potential.
2. Use of any medications (prescription or over-the-counter [OTC]) within 14 days of study drug administration; the use of cyclosporine or tacrolimus drugs is prohibited within 30 days prior to dosing and the use of biological therapies including but not limited to anti-tumour necrosis factor or anti-interleukin-6 drugs is prohibited within 60 days prior to dosing. An exception is made for limited amounts of paracetamol (acetaminophen) (up to a maximum of 4 g/ day) or ibuprofen (up to 1.2 g/day); the extent of nonsteroidal anti-inflammatory drug self-medication will be documented. Other exceptions will only be made if the rationale is clearly documented by the Investigator.
3. Current use of any vitamins or herbal supplements.
4. Use of hormone replacement therapy, oral contraceptives, intrauterine hormonal contraception within 30 days of screening, or injectable hormonal contraception within 3 months of screening.
5. Any vaccination with vaccines will be prohibited during study as well as within 30 days prior to (first) dosing in the study and within 30 days after the follow up visit.
6. History of drug/chemical/alcohol abuse within 6 months prior to Screening. History of alcohol consumption of > 21 units per week for males and > 14 units per week for females within 6 months prior to Check-in. In addition, no alcohol to be consumed within 24 hours of screening or Check-in. One unit of alcohol equals 1 pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
7. Positive alcohol breath test result or positive urine drug screen at Screening or Check-in.
8. Consumption of excessive xanthine (e.g. more than 8 cups of coffee or equivalent per day) within 1 month prior to screening.
9. History of serious bacterial, viral, fungal, or parasitic infection, including but not limited to viral hepatitis (hepatitis B or C or hepatitis caused by cytomegalovirus [CMV] or Epstein-Barr virus [EBV]), tuberculosis or Toxoplasma (T.) gondii in the past 5 years.
10. History of varicella zoster (chicken pox) or herpes zoster (shingles) in the past 5 years.
11. History of known or suspected immunodeficiency state or condition that would compromise the participant's immune status, or any factor that would pre-dispose the participant to develop an infection, including but not limited to human immunodeficiency virus (HIV).
12. Positive test for SARS-CoV-2 at Check-in.
13. Recent or ongoing infection, such as current evidence of ongoing or acute infection, history of repeated, chronic or opportunistic infections (e.g., recurrent folliculitis, other cutaneous infections or repeated pneumonia) or history of a serious bacterial infection within 6 months prior to dosing.
14. Positive hepatitis panel as defined by positive Hepatitis B surface antigen, Hepatitis B core antibody, or Hepatitis C antibody.
15. History of anaemia or any known or suspected condition that could be complicated by anaemia, or pre-dispose a participant to anaemia. Volunteers who have a history of iron deficiency anaemia for which a cause was identified and known not to be an ongoing concern (e.g. single episode of blood loss) and whose iron stores have fully recovered may be included. Participants will be excluded if haemoglobin is less than 12 g/dL.
16. ECG abnormalities in the resting ECG defined as:

    1. A corrected QT interval by Fredericia (QTcF) >450 msec for males and QTcF > 470 for females;
    2. QRS >120 msec;
    3. Personal or family history of congenital long QT syndrome or sudden death;
    4. ECG with QRS and/or T wave judged to be unfavourable for a consistently accurate QT measurement (e.g., neuromuscular artefact that cannot be readily eliminated, arrhythmias, indistinct QRS onset, low amplitude T wave, merged T- and U-waves, prominent U-waves);
    5. Evidence of atrial fibrillation, atrial flutter, complete branch block, Wolf-Parkinson-White Syndrome, or cardiac pacemaker.
17. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 1.5 times the upper limit of normal at Screening or Check-in.
18. Use of more than 5 cigarettes/day (or equivalent amount of chewing tobacco, e-cigarettes or nicotine patches) after Screening until Check-in. No smoking is allowed during confinement.
19. Have participated in another clinical trial within 3 months prior to screening.
20. Have donated blood within 4 weeks prior to screening.
21. Not willing and/or unable to consume investigational product that contains bovine and/or porcine products, or has a known or suspected allergy or hypersensitivity to bovine and/or porcine products.
22. Evidence of any active or chronic disease or condition that could interfere with, or which the treatment of the disease might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the Investigator (following a detailed medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory parameters). This includes a history or presence of any disease (e.g. malignancy), condition, or surgery (e.g., cholecystectomy or stomach operation) likely to affect drug absorption, distribution, metabolism, or excretion. Minor deviations of laboratory values from the normal range may be accepted, if judged by the Investigator as clinically irrelevant.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Adverse event assessed by Safety review committee | approximately not less than 1 month
  reported SAEs and AEs

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Opipari, MD, PhD, Study Chair — Odyssey Therapeutics
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No